CLINICAL TRIAL: NCT04966845
Title: The Effect of Surgical Face Mask on Exhaled Carbon Monoxide for Smokers During the COVID-19 Era.
Brief Title: Effect of Face Mask on Exhaled Carbon Monoxide of Smokers
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Professor of Cardiology, University of Athens
Other Study IDs: ExhaledCO
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Concentration of Exhaled Carbon Monoxide
Keywords: smoking; heat-not-burn cigarette; face mask; Carbon Monoxide
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Smokers: Exclusive smokers of conventional cigarettes
  Interventions: Diagnostic Test: measurement of concentration on exhaled Carbon Monoxide
- HNBC: Exclusive smokers of Heat-Not-Burn Cigarettes (HNBC)
  Interventions: Diagnostic Test: measurement of concentration on exhaled Carbon Monoxide
- Nonsmokers: Subjects that abstain from smoking for at least one year
  Interventions: Diagnostic Test: measurement of concentration on exhaled Carbon Monoxide

INTERVENTIONS:
Diagnostic Test: measurement of concentration on exhaled Carbon Monoxide — exhaled carbon monoxide (eCO) concentration [parts per million (ppm) was measured by a specific device [Bedfont Scientific, Maidstone, Kent UK]

SUMMARY:
Study of 120 healthy subjects without cardiovascular disease, 40 smokers of conventional cigarettes, 40 exclusive users of Heat-non-Burn Cigarettes and 40 nonsmokers.

Baseline measurements of CO will be performed in the morning after awakening without the use of any mask when they arrive at hospital. This time point is selected to detect the lowest exhaled CO levels after the abstinence of smoking during the sleep.

After baseline CO measurement, subjects will be randomly assigned to assess exhaled CO concentration at the end of an 8h morning shift wearing a mask at hospital, or to CO assessment at the end of an 8h morning period without mask out of the hospital (usually home stay). Then the subjects will be crossed over to CO assessment at end of an 8h period without mask out of the hospital after their shift or to an 8h afternoon period wearing a mask during an afternoon hospital shift respectively.

DETAILED DESCRIPTION:
Study of 120 healthy subjects without cardiovascular disease, 40 smokers of conventional cigarettes, 40 exclusive users of Heat-non-Burn Cigarettes and 40 nonsmokers.

All subjects are civil medical personnel working for the National Health System, in a Tertiary University Hospital in Athens. Also, working in a hospital environment will ensure the use of a mask during the shift.

Baseline measurements of CO will be performed in the morning after awakening without the use of any mask when they arrived at hospital. This time point is selected to detect the lowest exhaled CO levels after the abstinence of smoking during the sleep. CO has a half-life of 5-6 hours and consequently CO levels after the period of sleep (almost 8 hours) verge to decline or to normalize.

After baseline CO measurement, subjects will be randomly assigned to assess exhaled CO concentration at the end of an 8h morning shift wearing a mask at hospital, or to CO assessment at the end of an 8h morning period without mask out of the hospital (usually home stay). Then the subjects will be crossed over to CO assessment at end of an 8h period without mask out of the hospital after their shift or to an 8h afternoon period wearing a mask during an afternoon hospital shift respectively.

Measurements with and without mask will be done one hour after smoking the last cigarette. Subjects are inducted to smoke the same number of cigarettes or heats during their shift while wearing the mask as well as during the out-hospital period when not using a mask. During their shift they are instructed to wear the surgical mask constantly.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals without cardiovascular disease. 40 smokers of conventional cigarettes , 40 exclusive users of Heat-non-Burn Cigarettes and 40 nonsmokers.

Exclusion Criteria:

* i) abnormal renal function, ii) hepatic failure (bilirubin> 2 mg / dl), iii) active malignancy, iv) patients treated with drugs that affect platelet function, v) history of coronary artery disease or peripheral artery disease, vi) history of cardiomyopathy, vii) age<21 years old, viii) patients with thrombocytopenia (PLTs < 100x109/L), ix) anemia (HCT <28%), x) alcohol or drug abuse, xi) pregnancy, xii) risk factors for cardiovascular disease.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 120 healthy subjects without cardiovascular disease, 40 smokers of conventional cigarettes , 40 exclusive users of Heat-non-Burn Cigarettes and 40 nonsmokers. All subjects were civil medical personnel working for the National Health System, in a Tertiary University Hospital in Athens. They were all vaccinated and frequently tested for COVID-19. Also, working in a hospital environment ensured the use of a mask during the shift.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Change in exhaled CO levels with the use of surgical face mask | 8 hours
  ppm
Change in exhaled CO levels without the use of surgical face mask | 8 hours
  ppm

SECONDARY OUTCOMES:
Change in Aortic Elastic Properties with the use of surgical face mask | 8 hours
  Aortic elastic properties will be quantified by measuring Pulse Wave Velocity (m/sec), as assessed by a dedicated device(Mobil-O-Graph, IEM GmbH, Aachen, Germany)
Change in Aortic Elastic Properties with the use of surgical face mask | 8 hours
  Aortic elastic properties will be quantified by measuring augmentation index (%), as assessed by a dedicated device (Mobil-O-Graph, IEM GmbH, Aachen, Germany)
Change in Aortic Elastic Properties with the use of surgical face mask | 8 hours
  Aortic elastic properties will be quantified by measuring central blood pressure (mm Hg), as assessed by a dedicated device (Mobil-O-Graph, IEM GmbH, Aachen, Germany)
Change in Aortic Elastic Properties without the use of surgical face mask | 8 hours
  Aortic elastic properties will be quantified by measuring Pulse Wave Velocity (m/sec), as assessed by a dedicated device (Mobil-O-Graph, IEM GmbH, Aachen, Germany).
Change in Aortic Elastic Properties without the use of surgical face mask | 8 hours
  Aortic elastic properties will be quantified by measuring augmentation index (%), as assessed by a dedicated device (Mobil-O-Graph, IEM GmbH, Aachen, Germany).
Change in Aortic Elastic Properties without the use of surgical face mask | 8 hours
  Aortic elastic properties will be quantified by measuring central blood pressure (mm Hg), as assessed by a dedicated device (Mobil-O-Graph, IEM GmbH, Aachen, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, Professor, Principal Investigator — National and Kapodistrian University of Athens
Locations (2):
- Greece (2):
  - Konstantinos Katogiannis, Athens, Attica
  - "Attikon" University General Hospital, Athens, Attica

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ikonomidis I, Katogiannis K, Kourea K, Gavriella K, Tsilivarakis D, Lambadiari V, Kouretas D, Biondi-Zoccai G. The effect of smoking on exhaled carbon monoxide and arterial elasticity during prolonged surgical mask use in the COVID-19 era. Eur J Prev Cardiol. 2022 Nov 15;29(16):e355-e358. doi: 10.1093/eurjpc/zwac101. No abstract available. PMID 35798027